CLINICAL TRIAL: NCT03216876
Title: An Open-Label Study Of Ursolic Acid For Primary Sclerosing Cholangitis
Brief Title: A Study Of Ursolic Acid For Primary Sclerosing Cholangitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-001
Record Dates: First submitted 2016-01-05; First posted 2017-07-13 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Ursolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (Experimental): Healthy subjects will assigned to ursolic acid taken orally as a single dose of 40 mg, 80 mg, and 120 mg
  Interventions: Drug: Ursolic acid
- PSC Single Dose (Experimental): PSC subjects will assigned to ursolic acid taken orally as a single dose of 40 mg, 80 mg, and 120 mg
  Interventions: Drug: Ursolic acid
- PSC Multiple Dose (Experimental): PSC subjects assigned to treatment with daily oral ursolic acid at the dose determined to be optimal in the first phase of the study. The treatment will last for 24 weeks with an off-treatment follow up of 28 weeks
  Interventions: Drug: Ursolic acid

INTERVENTIONS:
Drug: Ursolic acid — Ursolic acid (UA) is a natural triterpenoid carboxylic acid, which has been studied for its anti-proliferative and anti-inflammatory activities.
  Other Names: urson; prunol; malol; 3-beta-3-hydroxy-urs-12-ene-28-oic-acid

SUMMARY:
This is an open-label, active treatment trial to determine the pharmacokinetics of orally administered ursolic acid and to assess the potential efficacy and safety of ursolic acid in subjects with primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
In the first phase of this trial, 6 healthy subjects and 2 PSC subjects will assigned to ursolic acid taken orally as a single dose of 40 mg, 80 mg, and 120 mg to determine the optimal dose in humans.

The second phase of this trial will involve 20 PSC subjects assigned to treatment with daily oral ursolic acid at the dose determined to be optimal in the first phase of the study. The treatment will last for 24 weeks with an off-treatment follow up of 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 - 70 years of age
* PSC documented by typically cholangiogram findings of strictures and dilations with no evidence of a secondary cause of sclerosing cholangitis
* Serum alkaline phosphatase greater than 1.5 times the upper limit of the normal reference range at the UC Davis Health Systems Clinical Laboratory
* AST and ALT ≤ 10 x ULN
* Serum creatinine < 2.0 mg/dL
* Mayo Activity Index of < 2 (in those with ulcerative colitis or Crohn's colitis)
* Negative serum pregnancy test for female subjects of childbearing potential, agreement to use a highly effective method of contraception during heterosexual intercourse (females of childbearing potential), lactating females must agree to discontinue nursing before starting study treatment, and barrier contraception during heterosexual intercourse (males not vasectomized).

Exclusion Criteria:

* Pregnancy
* Hepatic decompensation defined as ascites (or use of diuretics), episodes of hepatic encephalopathy, variceal bleeding or an INR > 1.2
* Positive HCV RNA or HBsAg, positive anti-mitochondrial antibody, alcohol consumption greater than 21oz/week for males or 14oz/week for females
* Clinically significant cardiac disease, history of cholangiocarcinoma, history of liver transplantation, history of cancers, other than non-melanomatous skin cancer, within 5 years prior to screening
* Ascending cholangitis within 60 days of screening
* Use of immunosuppressants including 6-mercaptopurine, azathioprine, methotrexate, mycophenolate mofetil, tacrolimus, cyclosporine, and anti-TNF or other biologics within 6 months of enrollment
* Use of antibiotics including vancomycin, metronidazole, or rifaximin within 60 days of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 hours
  Number of serious adverse events or Grade 3-4 biochemical abnormalities

SECONDARY OUTCOMES:
maximum plasma concentration (C¬max) | 24 hours
  Measured in mass of drug/ volume of fluid, The peak plasma concentration of a drug after administration.
half-life (t1/2), | 24 hours
  measured in time ,Time to reach Cmax.
volume of distribution (Vd) | 24 hours
  Measured in volume, The apparent volume in which a drug is distributed (i.e., the parameter relating drug concentration to drug amount in the body).
clearance | 24 hours
  Measured in Volume/ time, The volume of plasma cleared of the drug per unit time
Area under the concentration-time curve (AUC) | 24 hours
  Measured in mass/(volume*time), The integral of the concentration-time curve (after a single dose or in steady state).
Alanine aminotransferase (ALT) | 24 weeks
  Change in ALT from baseline to 24 weeks
Total bilirubin | 24 weks
  Change in total bilirubin from baseline to 24 weeks.
C-reactive Protein (CRP) | 24 weks
  Change in CRP from baseline to 24 weeks.
Mayo Risk Score (MRS) | 24 weks
  Change in MRS from baseline to 24 weeks.
Biochemical response | 24 weeks
  Reduction in serum alkaline phosphatase by 50% or to within the normal reference range and change in alkaline phosphatase from day 0 to week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowlus, MD, Principal Investigator — University of California, Davis
Locations (1):
- Univeristy of California Davis Medical Center, Sacramento, California, United States